CLINICAL TRIAL: NCT06777147
Title: Reproductive Health Outcomes in Young Patients with Ovarian Cancer After Surgical Treatment: a Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Raed Abdeltawab gomaa Selim, Dr, Assiut University
Other Study IDs: Ovarian cancer
Record Dates: First submitted 2024-12-22; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ovarian cancer (OC) is the second commonest gynecological cancer with an overall incidence of 1.4% , associated with high mortality rate , There are three major types of ovarian cancers: epithelial ovarian carcinomas, germ cell tumors, and stromal cell tumors .

Ovarian cancer directly affects fertility, as treatment consists of surgical removal of the reproductive system and/or exposure to gonadotoxic agents. However, patients in early stages who meet established criteria can be treated with fertility-sparing surgeries and reach equivalent oncological results to those of traditional treatments. Fertility preservation techniques such as cryopreservation of oocytes, embryos and ovarian tissue may also be offered in some situations.

Ovarian cancer (OC) has a high mortality rate and usually presents late in advanced stage, which poses challenges to management. Better understanding of the disease biology and application of radical surgery (RS) to achieve no visible residual tumor, alongside with chemotherapy, may lead to longer survival amongst these patients. Our purpose is to find out the fertility and survival rates of women with Overian Cancer in reproductive women who underwent surgical intervention. Radical Surgery for Overian cancer is one of the most challenging procedures in gynecologic oncology surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Women in reproductive age 18-45 yrs
2. Localized ovarian cancer
3. Patients undergoing surgical intervention

Exclusion Criteria:

1- Patients who refuse to participate in the study. 2 - children and manupausl women 3 - Diffuse peritoneal ,enteric and mesenteric disease or very poor patient 's performance status 4 -Patients who were treated with chemotherapy only and not operated

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Reproductive age Women ( >18yrs: 45yrs ) with Ovarian Cancers who had surgical intervention between 2020 : 2023
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of fertility rate of Reproductive age Women with Ovarian Cancer who underwent surgical intervention | From enrollment till the end of the study

SECONDARY OUTCOMES:
Morbidity and mortality | From enrollment till the end of the study
Sexual health | From enrollment till the end of the study

REFERENCES:
- [Background] Bhopal RS, Bansal N, Steiner M, Brewster DH; Scottish Health and Ethnicity Linkage Study. Does the 'Scottish effect' apply to all ethnic groups? All-cancer, lung, colorectal, breast and prostate cancer in the Scottish Health and Ethnicity Linkage Cohort Study. BMJ Open. 2012 Sep 25;2(5):e001957. doi: 10.1136/bmjopen-2012-001957. Print 2012. PMID 23012329
- [Background] Derlatka P, Sienko J, Grabowska-Derlatka L, Palczewski P, Danska-Bidzinska A, Bidzinski M, Czajkowski K. Results of optimal debulking surgery with bowel resection in patients with advanced ovarian cancer. World J Surg Oncol. 2016 Feb 29;14:58. doi: 10.1186/s12957-016-0800-1. PMID 26923029
- [Background] Chi DS, Eisenhauer EL, Lang J, Huh J, Haddad L, Abu-Rustum NR, Sonoda Y, Levine DA, Hensley M, Barakat RR. What is the optimal goal of primary cytoreductive surgery for bulky stage IIIC epithelial ovarian carcinoma (EOC)? Gynecol Oncol. 2006 Nov;103(2):559-64. doi: 10.1016/j.ygyno.2006.03.051. Epub 2006 May 22. PMID 16714056
- [Background] van de Laar R, IntHout J, Van Gorp T, Verdonschot S, van Altena AM, Gerestein CG, Massuger LF, Zusterzeel PL, Kruitwagen RF. External validation of three prognostic models for overall survival in patients with advanced-stage epithelial ovarian cancer. Br J Cancer. 2014 Jan 7;110(1):42-8. doi: 10.1038/bjc.2013.717. Epub 2013 Nov 19. PMID 24253502
- [Background] Patankar S, Burke WM, Hou JY, Tergas AI, Huang Y, Ananth CV, Neugut AI, Hershman DL, Wright JD. Risk stratification and outcomes of women undergoing surgery for ovarian cancer. Gynecol Oncol. 2015 Jul;138(1):62-9. doi: 10.1016/j.ygyno.2015.04.037. Epub 2015 May 11. PMID 25976399
- [Background] Chiva L, Lapuente F, Castellanos T, Alonso S, Gonzalez-Martin A. What Should We Expect After a Complete Cytoreduction at the Time of Interval or Primary Debulking Surgery in Advanced Ovarian Cancer? Ann Surg Oncol. 2016 May;23(5):1666-73. doi: 10.1245/s10434-015-5051-9. Epub 2015 Dec 29. PMID 26714955
- [Background] Rutten MJ, Boldingh JH, Schuit E, Trum H, van Driel W, Mol BW, Kenter GG, Buist MR. Development and internal validation of a prognostic model for survival after debulking surgery for epithelial ovarian cancer. Gynecol Oncol. 2014 Oct;135(1):13-8. doi: 10.1016/j.ygyno.2014.07.099. Epub 2014 Aug 2. PMID 25093289